CLINICAL TRIAL: NCT03166618
Title: A Multicenter, Single-Blind, Randomized, Parallel-Group, Controlled Study of the Safety and Effectiveness of JUVÉDERM VOLUMA® XC Injectable Gel for Correction of Temple Hollowing
Brief Title: Safety and Effectiveness of JUVÉDERM VOLUMA® XC Injectable Gel for Correction of Temple Hollowing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to stop the program.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VOLUMA-007
Record Dates: First submitted 2017-03-06; First posted 2017-05-25 (Actual); Results first posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Temple Hollowing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- VOLUMA® XC Treatment (Experimental): Participants will be treated with JUVÉDERM® VOLUMA® XC injectable gel in both temples (area above the eye). Participants are eligible for touch-up treatment 30 days later.
  Interventions: Device: Juvéderm® VOLUMA XC
- Control_No Treatment (No Intervention): No treatment is administered.

INTERVENTIONS:
Device: Juvéderm® VOLUMA XC — Juvéderm® VOLUMA XC hyaluronic acid injectable gel
  Arms: VOLUMA® XC Treatment

SUMMARY:
This study will evaluate the safety and effectiveness of JUVÉDERM VOLUMA XC injectable gel in adult participants seeking correction of temple hollowing.

ELIGIBILITY:
Inclusion Criteria:

-Has temple hollowing and is seeking restoration in the temple area.

Exclusion Criteria:

* Has temple hollowing due to due to trauma, congenital malformations, or lipodystrophy
* Has received permanent facial implants in the face or neck
* Has undergone fat injections
* Has tattoos, piercings, facial hair or scars that would interfere with visual assessment of the temple
* Has undergone semipermanent dermal filler treatment in the temple or mid-face within the past 36 months
* Has undergone dermal filler injections above the subnasale within the past 24 months
* Has temporal arteritis or history of temporal arteritis
* Has temporomandibular joint dysfunction
* Has eye inflammation or infection
* Has a history of detached retina, retinal vascular occlusion, narrow angle glaucoma, or neovascular eye disease
* Has ever received a facelift, browlift, or facial reconstructive surgery
* Has undergone mesotherapy or cosmetic treatment (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, liposuction, lipolysis, or other ablative procedures) anywhere in the face or neck or botulinum toxin injections within the past 6 months
* Has experienced trauma to the temple within the past 6 months or has residual deficiencies, deformities, or scarring
* Has a tendency to develop hypertrophic scarring
* Has a history of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), hyaluronic acid products, or Streptococcal protein
* Has porphyria or untreated epilepsy
* Has active autoimmune disease
* Has current cutaneous or mucosal inflammatory or infectious processes
* Is on a lidocaine, anticoagulation therapy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Amaratunge, Study Director — Allergan
Locations (1):
- Skin Care and Laser Physicians of Beverly Hills, Los Angeles, California, United States

REFERENCES:
- See also: More Information — http://allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Up to 189 subjects were planned; 1 subject was enrolled but did not receive treatment.
Period: Overall Study
Arm/Group | VOLUMA® XC Treatment | Control_No Treatment
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Study was Terminated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Up to 189 subjects were planned; 1 subject was enrolled in the control_No Treatment arm. Due to confidentiality considerations, baseline data is not being provided to protect participant privacy.
Groups:
- Total: Total of all reporting groups
Arm/Group | VOLUMA® XC Treatment | Control_No Treatment | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [unit: Participants]
Sex: Female, Male [unit: participants]
Ethnicity (NIH/OMB) [unit: Participants]
Race (NIH/OMB) [unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 1-Point Improvement (Decrease) in Both Temples as Assessed by the Evaluating Investigator Using the Allergan Temple Hollowing Scale (ATHS)
Description: The Evaluating Investigator will assess the participant's temple hollowing using the ATHS 5-point scale where: 0=convex, rounded temple to 4=severe, deeply recessed, sunken appearance. A 1-point decrease from Baseline indicates improvement.
Time Frame: Change from Baseline to Month 3
Population: Up to 189 subjects were planned; 1 subject was enrolled in the control_No Treatment arm. Terminated study; no treatment was administered and no analyses were conducted.
Arm/Group | VOLUMA® XC Treatment | Control_No Treatment
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants "Improved" or "Much Improved" as Assessed by the Evaluating Investigator Using the Global Aesthetic Improvement Scale (GAIS)
Description: The Evaluating Investigator will assess the participant's temple area using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. The percentage of participants who the Evaluating Investigator assesses as 2=much improved or 1=improved will be reported.
Time Frame: Month 3
Population: as for outcome 1
Arm/Group | VOLUMA® XC Treatment | Control_No Treatment
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants "Improved" or "Much Improved" as Assessed by the Participant Using the GAIS
Description: The participant will assess their temple area using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. The percentage of participants who assess themselves as 2=much improved or 1=improved will be reported.
Time Frame: Month 3
Population: as for outcome 1
Arm/Group | VOLUMA® XC Treatment | Control_No Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Up to 189 subjects were planned; 1 subject was enrolled in the control_No Treatment arm
Arm/Group | VOLUMA® XC Treatment | Control_No Treatment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Due to low patient enrollment, the target number of participants needed to achieve target power and statistically reliable results was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The TI is responsible for compliance with the protocol at the investigational site. A representative of Allergan will make frequent contact with the TI and his/her research staff and will conduct regular monitoring visits at the site to review subject and device accountability records for compliance with the protocol

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT03166618/Prot_SAP_000.pdf